CLINICAL TRIAL: NCT03352518
Title: Performance Characteristics and Safety Assessment of a Non-invasive Glucose Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-12-02
Record Dates: First submitted 2017-11-13; First posted 2017-11-24 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMD data collection (Experimental): Subjects will intensively collect spectral raman data in a home-based setting for 5 days using WM3.4NR and comparators.
  Interventions: Device: WM3.4NR

INTERVENTIONS:
Device: WM3.4NR — The investigational medical device will collect spectral raman data from tissue.

SUMMARY:
This clinical study has been launched to collect spectral raman data paired with validated glucose reference values in private homes of subjects.

DETAILED DESCRIPTION:
Subjects will collect spectral raman data on device every 15 minutes for 10 hours a day for five days. The five days will be distributes with in a timeframe of ten days. A Flash Glucose Monitor will be used as a comparator. In addition to this, four daily capillary Blood Glucose readings will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older
* Diabetic patients (all types)

Exclusion Criteria:

* Pregnant women
* Subjects not able to understand and read Danish
* In investigator's opinion, subject is not able to follow instructions as specified in the protocol
* Subjects not able to hold hand/arm steadily
* Extensive skin changes, tattoos or diseases on probe application site
* Known allergy to medical grade alcohol used to disinfect skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Generation and validation of predictive calibration models | 3 months
  The collected data will generate individual calibration models capable of predicting tissue glucose concentrations. An evaluation of the models by the consensus error grid will be performed.

SECONDARY OUTCOMES:
Safety assessment of the intervention by the paucity of adverse events | 3 months
  The number of subjects experiencing device-related adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, Principal Investigator — University Hospital Odense
Locations (1):
- Department of Endocrinology M, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No